CLINICAL TRIAL: NCT04871321
Title: Discovery of Molecular Biomarkers for Predicting Response Through RNA Sequencing in Patients With Advanced Biliary Tract Cancer Who Received Nab-paclitaxel Plus Gemcitabine-cisplatin
Brief Title: Biomarker Discovery in Patients With Advanced Biliary Tract Cancer
Status: Completed | Type: Observational
Sponsor: CHA University (Other)
Collaborators: Dong-A Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-03-045
Record Dates: First submitted 2021-04-26; First posted 2021-05-04 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Biliary Tract Cancer; Cholangiocarcinoma; Gallbladder Cancer
Keywords: Biliary Tract cancer; Gemcitabine; Cisplatin; nab-paclitaxel; RNA sequencing; biomarker
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Immunohistochemistry; Base Sequence; Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Tissue, Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gem/Cis/nab-P: Gemcitabine + Cisplatin + Nab-Paciltaxel
  Interventions: Drug: nab-paclitaxel plus gemcitabine-cisplatin

INTERVENTIONS:
Drug: nab-paclitaxel plus gemcitabine-cisplatin — - gemcitabine 800mg/m2 + cisplatin 25 mg/m2 + nab-paclitaxel 100mg/m2 on day 1 and day 8, every 21 days
  Other Names: immunohistochemistry, NGS, RNA-sequencing, Liquid biopsy

SUMMARY:
Biliary tract cancer is a rare gastrointestinal malignant neoplasm and includes intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gall bladder cancer. Curative surgical resection offers the only chance for cure. However, most patients with BTC are diagnosed at an unresectable stage. Therefore, the survival outcomes of patients with advanced biliary tract cancer remain dismal.

The combination of gemcitabine and cisplatin has become the current standard for advanced BTCs since the landmark ABC-02 trial in 2010. However, the median overall survival of Gem/Cis chemotherapy is less than 1 year. Recently, a triplet regimen of gemcitabine, cisplatin, and nab-paclitaxel showed promising results in a single-arm phase II multicenter study.

However, biliary tract cancer is a group of heterogenous diseases by site and genetic alteration, and this diversity may lead differences in response to systemic chemotherapy.

Transcriptome analysis through RNA-sequencing has rarely been performed in advanced biliary tract cancer, and even if it has performed, only small number of patients were included. Further research on multi-omics data is needed on the necessity and clinical significance in treatment of biliary tract cancer.

DETAILED DESCRIPTION:
Using biopsy specimen (formalin fixed paraffin embedded tissue), in-house NGS and RNA-sequencing will be performed simultaneously. Through this, investigators will discover biomarkers based on multi-omics data that predict response to systemic chemotherapy (nab-paclitaxel plus gemcitabine-cisplatin). In addition, blood sampling will be performed in parallel to conduct research on cell-free DNA and circulating tumor cell analysis related to response and progression on chemotherapy; before administration of chemotherapy, 3 months after chemotherapy, 6 months after chemotherapy, the time of disease progression (if possible), before curative resection (if possible).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years old
* Capable of understanding and complying with the protocol requirements and signed informed consent
* The patients were confirmed as bilary tract cancer (gall bladder cancer, extrahepatic cholangiocarcinoma, intrahepatic cholangiocarcinoma) by histopathology or cytology
* Patients with inoperable or metastatic or recurrent biliary tract cancer
* Patients who underwent in-house next-generation sequencing
* Patients planning to receive Gemcitabine, Cisplatin, nab-paclitaxel triplet chemotherapy
* At least one measurable objective lesion was identified based on the RECIST 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* The expected survival a ≥3 months

Exclusion Criteria:

* The subject has uncontrolled, significant intercurrent or recent illness including infection for organ failure
* Prior palliative chemotherapy for biliary tract cancer
* Dementia, altered mental state, or any mental illness that prevents understanding or informed consent
* Other conditions that researchers not think to be suitable for enrollment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced biliary tract cancer will be recruited at CHA Bundang Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
collected tumor samples | through study completion, an average of 2 years
  tumor samples from patients with hepatobiliary cancers (incidence of genetic alteration, association with treatment response and survival duration)
collected blood samples | through study completion, an average of 2 years
  blood samples from patients with hepatobiliary cancers (incidence of genetic alteration, association with treatment response and survival duration)

SECONDARY OUTCOMES:
Multi-omics analysis | 2 years
  Multi-omics analysis to further subtype and find therapeutic targets of biliary tract cancer
Biomarkers on the efficacy of Gemcitabine/Cisplatin/Nab-paclitaxel for advanced biliary tract cancer | 2 years
  Molecular biomarker associated with overall survival, progression-free survival and objective response rate in patients who receive Gemcitabine/Cisplatin/Nab-paclitaxel chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Hongjae Chon, MD,PhD, Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jarnagin WR, Fong Y, DeMatteo RP, Gonen M, Burke EC, Bodniewicz BS J, Youssef BA M, Klimstra D, Blumgart LH. Staging, resectability, and outcome in 225 patients with hilar cholangiocarcinoma. Ann Surg. 2001 Oct;234(4):507-17; discussion 517-9. doi: 10.1097/00000658-200110000-00010. PMID 11573044
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Kim BJ, Hyung J, Yoo C, Kim KP, Park SJ, Lee SS, Park DH, Song TJ, Seo DW, Lee SK, Kim MH, Park JH, Cho H, Ryoo BY, Chang HM. Prognostic factors in patients with advanced biliary tract cancer treated with first-line gemcitabine plus cisplatin: retrospective analysis of 740 patients. Cancer Chemother Pharmacol. 2017 Jul;80(1):209-215. doi: 10.1007/s00280-017-3353-2. Epub 2017 Jun 8. PMID 28597043
- [Background] Shroff RT, Javle MM, Xiao L, Kaseb AO, Varadhachary GR, Wolff RA, Raghav KPS, Iwasaki M, Masci P, Ramanathan RK, Ahn DH, Bekaii-Saab TS, Borad MJ. Gemcitabine, Cisplatin, and nab-Paclitaxel for the Treatment of Advanced Biliary Tract Cancers: A Phase 2 Clinical Trial. JAMA Oncol. 2019 Jun 1;5(6):824-830. doi: 10.1001/jamaoncol.2019.0270. PMID 30998813
- [Background] Chae H, Kim D, Yoo C, Kim KP, Jeong JH, Chang HM, Lee SS, Park DH, Song TJ, Hwang S, Kim KH, Song GW, Ahn CS, Lee JH, Hwang DW, Kim SC, Jang SJ, Hong SM, Kim TW, Ryoo BY. Therapeutic relevance of targeted sequencing in management of patients with advanced biliary tract cancer: DNA damage repair gene mutations as a predictive biomarker. Eur J Cancer. 2019 Oct;120:31-39. doi: 10.1016/j.ejca.2019.07.022. Epub 2019 Aug 30. PMID 31476489
- [Background] Nakamura H, Arai Y, Totoki Y, Shirota T, Elzawahry A, Kato M, Hama N, Hosoda F, Urushidate T, Ohashi S, Hiraoka N, Ojima H, Shimada K, Okusaka T, Kosuge T, Miyagawa S, Shibata T. Genomic spectra of biliary tract cancer. Nat Genet. 2015 Sep;47(9):1003-10. doi: 10.1038/ng.3375. Epub 2015 Aug 10. PMID 26258846
- [Background] Chu KJ, Ma YS, Jiang XH, Wu TM, Wu ZJ, Li ZZ, Wang JH, Gao QX, Yi B, Shi Y, Wang HM, Gu LP, Zhang SQ, Wang GR, Liu JB, Fu D, Jiang XQ. Whole-Transcriptome Sequencing Identifies Key Differentially Expressed mRNAs, miRNAs, lncRNAs, and circRNAs Associated with CHOL. Mol Ther Nucleic Acids. 2020 Sep 4;21:592-603. doi: 10.1016/j.omtn.2020.06.025. Epub 2020 Jun 27. PMID 32721879
- [Background] Cheon J, Lee CK, Sang YB, Choi HJ, Kim MH, Ji JH, Ko KH, Kwon CI, Kim DJ, Choi SH, Kim C, Kang B, Chon HJ. Real-world efficacy and safety of nab-paclitaxel plus gemcitabine-cisplatin in patients with advanced biliary tract cancers: a multicenter retrospective analysis. Ther Adv Med Oncol. 2021 Aug 7;13:17588359211035983. doi: 10.1177/17588359211035983. eCollection 2021. PMID 34394748